CLINICAL TRIAL: NCT02044926
Title: Intraductal Papillary Mucinous Neoplasm (IPMN) With Malignant Change: Prospective Study to Assess Diagnostic Performance of CT and Magnetic Resonance Imaging (MR) According to International Consensus Guidelines 2012
Brief Title: Intraductal Papillary Mucinous Neoplasm With Malignant Change
Status: Terminated | Type: Observational
Why Stopped: Because patient enrollment is so difficult.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jae Ho Byun, Jae Ho Byun, Asan Medical Center
Other Study IDs: S2013-1472-0002
Record Dates: First submitted 2014-01-21; First posted 2014-01-24 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: IPMN

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Purpose:

To investigate diagnostic performance of CT and MR in intraductal papillary mucinous neoplasm with malignant change according to international consensus guidelines 2012.

Hypothesis: According to 2012 consensus guidelines, enhanced solid component and main pancreatic duct size of larger than 10 mm will be significant.

DETAILED DESCRIPTION:
1. Purpose

   * To investigate diagnostic performance of CT and MR in intraductal papillary mucinous neoplasm with malignant change according to international consensus guidelines 2012
2. Enroll criteria

   * Patient who is suspected to have pancreas IPMN on imaging
   * Interval between imaging study and surgery is less than 2 months
   * Who is scheduled for surgery due to IPMN

ELIGIBILITY:
Inclusion Criteria:

* Patients who is suspected to have IPMN by imaging study or clinician
* Time interval between imaging study and surgery less than 2 months

Exclusion Criteria:

* Patients who have pathology results not by surgery
* Who is less than 20 years old
* Who cannot voluntarily agree study design

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patents who are suspected to have pancreas IPMN by clinicians or imaging studies
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Imaging predictor of malignant IPMN of the pancreas | one month
  We will assess baseline CT and MRI findings of patients within one month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ho Byun, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea